CLINICAL TRIAL: NCT02649556
Title: A 26-week Extension Study to Determine the Biological and Functional Changes in Healthy Smokers Who Switched From Conventional Cigarettes (CC) to Tobacco Heating System 2.2 (THS 2.2) Compared to Those Who Continued to Smoke CC in the ZRHR-ERS-09-US Study
Brief Title: A 26-week Extension of the ZRHR-ERS-09-US Study Evaluating Biological and Functional Changes in Healthy Smokers After Switching to THS 2.2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRHR-ERS-09-EXT-US; ZRHR-ERS-09-EXT-US (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking
Keywords: Modified risk tobacco product; Conventional cigarette; Exposure response; Smoking; Tobacco Heating System
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THS 2.2 (Experimental): Ad libitum use of THS 2.2
  Interventions: Other: THS 2.2
- CC (Active Comparator): Ad libitum use of CC
  Interventions: Other: CC

INTERVENTIONS:
Other: THS 2.2 — Ad libitum use of THS 2.2 in an ambulatory setting for 26 weeks.
  Arms: THS 2.2
Other: CC — Ad libitum use of CC in an ambulatory setting for 26 weeks.
  The subject's own preferred brands of CC (no brand restriction) continue to be used as the reference product.
  Arms: CC

SUMMARY:
The objective of the ZRHR-ERS-09-EXT-US study is to further assess the effect of the Tobacco Heating System 2.2 (THS 2.2), a candidate Modified Risk Tobacco Product, compared to conventional cigarettes (CC) on the components of the "smokers' health profile" for a prolonged period of 26 weeks, providing additional information to the results of the original study ZRHR-ERS-09-US of 26-week exposure (NCT02396381). In total, the ZRHR-ERS-09-EXT-US study will extend the exposure period to 52 weeks.

DETAILED DESCRIPTION:
The ZRHR-ERS-09-EXT-US study is a 26-week extension of the original study ZRHR-ERS-09-US.

The subjects in the Full Analysis Set - As Exposed (FAS-EX) included subjects for combined analyses from the original six month study (ZRHR-ERS-09-US ) who did not enter the extension study (ZRHR-ERS-09-EXT-US).

This study was conducted as a separate investigation, as a follow-up of the randomized exposure period of the original study, extending the exposure from Week 26 (Visit 10 [V10]) to Week 52 (Visit 16 [V16]), and using the same sites.

Subjects continued to use the product they were randomized to in the original study ZRHR-ERS-09-US (THS 2.2 arm or CC arm).

ELIGIBILITY:
Inclusion Criteria:

* Subject completed V10 of the original study (ZRHR-ERS-09-US).
* The subject is willing to comply to study procedures and to continue to use the product he/she was allocated to during the original study (THS 2.2 or CC) for an additional 26 weeks at V10.
* Subject has given written informed consent to enter the 26-week extension study at V10.

Exclusion Criteria:

* Clinically relevant medical conditions that in the opinion of the investigators would jeopardize the safety of the participant.
* As per judgment of the PI(s) or designee(s), the subject cannot participate in the study for any reason (e.g. medical, psychiatric and/or social reason).
* Subject has made an attempt to quit using tobacco-containing products (e.g. CC and THS 2.2) during the original study.
* Female subject is pregnant or breast feeding.
* Female subject who does not agree to use an acceptable method of effective contraception.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Danielle Armas, MD, Principal Investigator — Celerion Arizona; Leonard Dunn, MD, Principal Investigator — Clinical Research West Florida; Hugh Coleman, MD, Principal Investigator — Covance; George Stoica, MD, Principal Investigator — Compass Research; Mark Adams, MD, Principal Investigator — Central Kentucky Research Associate; Peter Davidson, MD, Principal Investigator — Celerion Lincoln; John Rubino, MD, Principal Investigator — PMG Research of Raleigh; George Raad, MD, Principal Investigator — PMG Research of Charlotte; Kevin Cannon, MD, Principal Investigator — PMG Research of Wilmington; Derek Schroder, MD, Principal Investigator — PMG Research of Cary; Stephanie Powell, MD, Principal Investigator — PMG Research of Bristol; William Smith, MD, Principal Investigator — NOCCR; Darrell Herrington, MD, Principal Investigator — Benchmark; Laurence Chu, MD, Principal Investigator — Benchmark; William Seger, MD, Principal Investigator — Benchmark; David Subich, MD, Principal Investigator — Compass Research; Lon Lynn, MD, Principal Investigator — Clinical Research West Florida; Isabel Kuhare-Arcure, MD, Principal Investigator — Midwest Clinical Research; Keith Scott, MD, Principal Investigator — National Clinical Research
Locations (19):
- United States (19):
  - Celerion Arizona, Tempe, Arizona
  - Clinical Research West Florida, Clearwater, Florida
  - Covance, Inc, Daytona Beach, Florida
  - Compass Research, Orlando, Florida
  - Clinical Research West Florida, Tampa, Florida
  - Compass Research, The Villages, Florida
  - Central Kentucky Research Associate, Lexington, Kentucky
  - Celerion Lincoln, Lincoln, Nebraska
  - PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Midwest Clinical Research, Dayton, Ohio
  - PMG Research of Bristol, Bristol, Tennessee
  - NOCCR, Knoxville, Tennessee
  - Benchmark, Austin, Texas
  - Benchmark, Fort Worth, Texas
  - Benchmark, San Angelo, Texas
  - National Clinical Research, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansari SM, Hession PS, David M, Blanc N, de La Bourdonnaye G, Pouly S, Haziza C. Impact of switching from cigarette smoking to tobacco heating system use on biomarkers of potential harm in a randomized trial. Biomarkers. 2024 Jul;29(5):298-314. doi: 10.1080/1354750X.2024.2358318. Epub 2024 Jun 7. PMID 38804903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 984 subjects (488 in the THS arm and 496 in the CC arm) who were enrolled and randomized into the original study, NCT02396381, 672 subjects were enrolled into the extension study (309 in the THS arm and 363 in the CC arm).
Pre-assignment Details: 672 subjects enrolled in the extension study; the 857 subjects in the Full Analysis Set - As Exposed (FAS-EX) included subjects for combined analyses from the original six month study who did not enter the extension study. The analysis was performed according to subjects' exposure over the 12 month period as detailed in "Arm/Group" (Reporting Groups) table.
Groups:
- THS 2.2 Use: This reporting group comprised 230 subjects. The "THS 2.2 use" product use category was defined as THS use of 70% or more over the entire analysis period. (≥1 THS 2.2 or CC, and ≥70% THS 2.2 use over the analysis period, and ≥70% THS 2.2 use on >50% of days in the analysis period.)
- CC Use: This reporting group comprised 424 subjects. The "CC use" product use category was defined as THS use of less than 1% over the entire analysis period. (≥1 THS 2.2 or CC use, and <1% THS 2.2 use over the entire analysis period and <1% THS 2.2 use on ≥ 50% of days in the analysis period.)
- Dual Use: This reporting group comprised 152 subjects. The "Dual use" product use category was defined as THS use of less than 70% over the entire analysis period. (≥ 1 THS 2.2 or CC and, 1% ≤THS 2.2 <70% over the analysis period, or THS 2.2-use and CC use categories do not apply to 50% of these days.)
- Other Use: This reporting group comprised 51 subjects. "Other use" refers to any other product use over the entire analysis period. (Subjects with missing product use data, subjects using e-cigarettes or other tobacco products, quitters, or subjects who switched across different use patterns.)
Period: Overall Study
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Started | 230 | 424 | 152 | 51
Completed | 167 | 312 | 102 | 28
Not Completed | 63 | 112 | 50 | 23

BASELINE CHARACTERISTICS:
Groups:
- THS 2.2 Use: The "THS 2.2 use" product use category was defined as THS use of 70% or more over the entire analysis period.
  (≥1 THS 2.2 or CC, and ≥70% THS 2.2 use over the analysis period, and ≥70% THS 2.2 use on >50% of days in the analysis period.)
- CC Use: The "CC use" product use category was defined as THS use of less than 1% over the entire analysis period.
  (≥1 THS 2.2 or CC use, and <1% THS 2.2 use over the entire analysis period and <1% THS 2.2 use on ≥ 50% of days in the analysis period.)
- Dual Use: The "Dual use" product use category was defined as THS use of less than 70% over the entire analysis period.
  (≥ 1 THS 2.2 or CC and, 1% ≤THS 2.2 <70% over the analysis period, or THS 2.2-use and CC use categories do not apply to 50% of these days.)
- Other Use: "Other use" refers to any other product use over the entire analysis period. (Subjects with missing product use data, subjects using e-cigarettes or other tobacco products, quitters, or subjects who switched across different use patterns.)
- Total: Total of all reporting groups
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use | Total
Number analyzed (Participants) | 230 | 424 | 152 | 51 | 857
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.68) | 45.2 (9.54) | 44.2 (9.76) | 44.5 (8.21) | 44.6 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 180 | 67 | 19 | 353
  Male | 143 | 244 | 85 | 32 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 28 | 6 | 2 | 53
  Not Hispanic or Latino | 213 | 396 | 146 | 49 | 804
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 2 | 1 | 6
  Asian | 2 | 5 | 0 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 3
  Black or African American | 41 | 73 | 25 | 12 | 151
  White | 182 | 338 | 123 | 36 | 679
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 1 | 10
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (4.06) | 27.1 (4.13) | 26.9 (4.25) | 26.6 (4.91) | 27.0 (4.18)

OUTCOME MEASURES:

1. Primary Outcome: Levels of High Density Lipoprotein C (HDL-C).
Description: Concentrations (mg/dL) measured in serum. Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: Full Analysis Set - As Exposed Analysis (FAS-EX). Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 168 | 315 | 103 | 28
mg/dL | 52.2 [49.5 to 54.8] | 50.6 [48.9 to 52.3] | 54.0 [49.7 to 58.4] | 54.7 [49.2 to 60.3]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of LS Mean difference of HDL-C levels between CC and THS 2.2 and related 95% CI; Test type: Other; LS Mean Difference = 1.75, 95% CI 2-sided [-0.160 to 3.65]; Mixed model conducted on original values with visit, baseline value and its interaction with visit, sex, Caucasian origin, product use pattern category and its interaction with visit, and other baseline covariates relevant for the specific clinical risk endpoint as fixed effect factors and site as a random effect

2. Primary Outcome: Levels of White Blood Cells (WBC).
Description: Total count in blood (GI/L). Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: GI/L
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 167 | 312 | 102 | 28
GI/L | 6.73 [6.47 to 6.99] | 7.31 [7.07 to 7.54] | 7.28 [6.85 to 7.71] | 7.57 [6.85 to 8.29]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of LS Mean difference of White Blood Cell counts between CC and THS 2.2 and related 95% CI; Test type: Other; LS Mean Difference = -0.413, 95% CI 2-sided [-0.694 to -0.131]; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1).
Description: FEV1 post-bronchodilator and expressed as percentage predicted (FEV1 %pred). Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent of predicted FEV1
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 153 | 288 | 95 | 27
Percent of predicted FEV1 | 93.2 [91.1 to 95.2] | 92.3 [90.7 to 94.0] | 91.1 [88.2 to 94.1] | 95.2 [90.1 to 100]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of LS Mean difference of FEV1 levels between CC and THS 2.2 and related 95% CI; Test type: Other; LS Mean Difference = 0.914, 95% CI 2-sided [-0.339 to 2.17]; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Concentrations of Soluble Intercellular Adhesion Molecule 1 (sICAM-1).
Description: Concentrations (ng/mL) measured in serum. Geometric Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 168 | 315 | 103 | 28
ng/mL | 246 [230 to 263] | 258 [244 to 272] | 269 [252 to 286] | 255 [222 to 292]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of relative reduction of sICAM-1 levels between CC and THS 2.2 and related 95% CI; Test type: Other; % Relative Reduction = 3.11, 95% CI 2-sided [0.0231 to 6.10] — Derived as 100 x (1 - Geometric LS Mean Ratio); Mixed model conducted on log-transformed values with visit, log-transformed baseline value and its interaction with visit, sex, Caucasian origin, product use pattern category and its interaction with visit, and other baseline covariates relevant for the specific clinical risk endpoint as fixed effect factors and site as a random effect

5. Primary Outcome: Concentrations of 11-dehydrothromboxane B2 (11-DTXB2).
Description: Concentrations measured in urine and expressed as concentration adjusted for creatinine (pg/mg creat). Geometric Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 166 | 312 | 102 | 27
pg/mg creat | 582 [518 to 654] | 586 [538 to 638] | 595 [510 to 693] | 536 [396 to 727]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of relative reduction of 11-DTXB2 levels between CC and THS 2.2 and related 95% CI; Test type: Other; % Relative Reduction = 3.44, 95% CI 2-sided [-8.74 to 14.3] — Derived as 100 x (1-Geometric LS Mean Ratio); [other analysis details as in outcome 4, analysis 1]

6. Primary Outcome: Concentrations of 8-epi-prostaglandin F2α (8-epi-PGF2α).
Description: as for outcome 5
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 167 | 312 | 102 | 27
pg/mg creat | 307 [279 to 338] | 327 [307 to 348] | 326 [293 to 362] | 364 [289 to 458]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of relative reduction of 8-epi-PGF2α levels between CC and THS 2.2 and related 95% CI; Test type: Other; % Relative Reduction = 7.15, 95% CI 2-sided [-1.03 to 14.7] — Derived as 100 x (1 - Geometric LS Mean Ratio); [other analysis details as in outcome 4, analysis 1]

7. Primary Outcome: Concentrations of Total 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (Total NNAL).
Description: as for outcome 5
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 167 | 312 | 102 | 27
pg/mg creat | 133 [105 to 168] | 269 [238 to 305] | 253 [207 to 309] | 304 [214 to 431]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of relative reduction of Total NNAL levels between CC and THS 2.2 and related 95% CI; Test type: Other; % Relative Reduction = 46.3, 95% CI 2-sided [36.2 to 54.8] — Derived as 100 x (1 - Geometric LS Mean Ratio); [other analysis details as in outcome 4, analysis 1]

8. Primary Outcome: Levels of Carboxyhemoglobin (COHb).
Description: Carboxyhemoglobin (COHb) is assayed from whole blood. Expressed as % of saturation of hemoglobin. Geometric Mean values are provided as descriptive statistics.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
Number analyzed (Participants) | 141 | 257 | 86 | 26
percent change | 2.59 [2.24 to 3.01] | 4.06 [3.77 to 4.38] | 3.92 [3.44 to 4.46] | 5.22 [4.47 to 6.11]
Statistical Analysis 1: Comparison: THS 2.2 Use vs CC Use; The analysis will determine the effect of THS 2.2 compared to CC at Month 12 on the components of the "smokers' health profile". This study has no formal pre-specified hypotheses associated with the study objectives. Estimates of THS 2.2 effect will be presented by mean of relative reduction of COHb levels between CC and THS 2.2 and related 95% CI; Test type: Other; % Relative Reduction = 31.7, 95% CI 2-sided [23.3 to 39.1] — Derived as 100 x (1 - Geometric LS Mean Ratio); [other analysis details as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 18 months (from March 2015 to September 2016)
Description: Of the 984 subjects who started the original study (NCT02396381), 20 subjects without a valid safety assessment and 24 subjects from a site terminated for non-GCP compliance were excluded from the safety population (N=940). The safety population comprised the 857 subjects of the Full Analysis Set - As Exposed (FAS-EX), who had at least one record of reported product use post randomization, and 83 subjects who were randomized and had at least 1 valid safety assessment.
Groups:
- Dual Use: The "Dual use" product use category was defined as THS use of less than 70% over the entire analysis period.
  (≥ 1 THS 2.2 or CC and, 1% ≤THS 2.2 <70% over the analysis period, or THS 2.2-use and CC use categories do not apply to 50% of these days.)
  .
Arm/Group | THS 2.2 Use | CC Use | Dual Use | Other Use
All-Cause Mortality (participants affected / at risk) | 1/241 | 1/434 | 0/159 | 1/106
Serious Adverse Events (participants affected / at risk) | 12/241 | 15/434 | 1/159 | 1/106
Other Adverse Events (participants affected / at risk) | 40/241 | 87/434 | 26/159 | 13/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Use (N=241) | CC Use (N=434) | Dual Use (N=159) | Other Use (N=106)
Appendicitis with Peritonitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis with Nephrolithiasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Head injury with Seizure (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture, Clavicle fracture, Pulmonary contusion, Pleural effusion, and Traumatic Hemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Alchohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Metastases to small intestine with Anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte with Cervical Myelopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bereavement and Adjustment Disorder with Depressed Mood (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THS 2.2 Use (N=241) | CC Use (N=434) | Dual Use (N=159) | Other Use (N=106)
Upper respiratory tract infection (Infections and infestations) | 21 (25) | 40 (45) | 11 (14) | 8 (9)
Hypertension (Vascular disorders) | 9 (13) | 26 (40) | 9 (11) | 4 (5)
Blood triglycerides increased (Investigations) | 10 (10) | 26 (28) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02649556/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT02649556/SAP_001.pdf